CLINICAL TRIAL: NCT03183141
Title: ECOSPOR IV: An Open-Label Extension of Study SERES-012 and Open-Label Program for Evaluating SER-109 in Subjects With Recurrent Clostridioides Difficile Infection (RCDI)
Brief Title: ECOSPOR IV: An Open-Label Study Evaluating SER-109 in Recurrent Clostridioides Difficile Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seres Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SERES-013
Expanded Access: NCT02437500 (Approved for marketing)
Record Dates: First submitted 2017-06-08; First posted 2017-06-09 (Actual); Results first posted 2023-03-31 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides infection; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Gram-Positive Bacterial Infections; Communicable Diseases
MeSH Terms: conditions — Clostridium Infections; Gastrointestinal Diseases; Digestive System Diseases; Intestinal Diseases; Gram-Positive Bacterial Infections; Communicable Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SER-109 (Experimental): Received oral dose of SER-109
  Interventions: Biological: SER-109

INTERVENTIONS:
Biological: SER-109 — SER-109, an oral, biologically derived, live microbiome therapeutic that comprises purified bacterial spores
  Other Names: Firmicutes spores

SUMMARY:
Cohort 1: Subjects who had a Clostridioides difficile infection (CDI) recurrence in study SERES-012 within 8 weeks of receipt of study drug will be eligible. The purpose of this cohort is to assess safety and efficacy of SER-109 in reducing recurrence of CDI in adults who had a CDI recurrence within 8 weeks after receipt of SER-109 or Placebo in study SERES-012.

Cohort 2: Cohort 2 is an open-label program for subjects who were not part of SERES-012. The purpose of this cohort is to describe safety and tolerability of SER-109 in subjects 18 years of age or older with at least a first recurrence of CDI.

DETAILED DESCRIPTION:
Cohort 1 is an open-label extension of study SERES-012. Subjects who had a CDI recurrence in study SERES-012 within 8 weeks of receipt of study drug, have responded to a course of standard of care (SOC) antibiotic treatment, will receive an oral dose of SER-109. A treatment regimen of SER-109 is defined as an oral dose of SER-109 (4 capsules once daily) for 3 consecutive days.

Approximately 30 eligible subjects with recurrent CDI disease from study SERES-012 are expected to enroll. Screening for this study will begin at the Recurrence Visit of Study SERES-012.

Cohort 2 is an open-label program for subjects who were not part of SERES-012. Subjects 18 years of age or older who had one or more CDI recurrence and have responded to a course of antibiotic treatment will receive an oral dose of SER-109. The CDI recurrence must be confirmed by a positive C. difficile stool toxin or polymerase chain reaction (PCR) assay to confirm eligibility. A treatment regimen of SER-109 is defined as an oral dose of SER-109 (4 capsules once daily) for 3 consecutive days.

Approximately 200 eligible subjects with recurrent CDI disease are expected to enroll.

ELIGIBILITY:
Cohort 1 Main Inclusion Criteria:

1. Previously enrolled in Study SERES-012, had CDI recurrence within 8 weeks after receipt of a treatment regimen of SER-109 or placebo
2. Signed informed consent prior to initiation of any study-specific procedure or treatment. The subject, or their legally authorized representative, must be able to provide written informed consent and understand the potential risks and benefits from study enrollment and treatment.
3. The CDI recurrence in Study SERES-012 must have met the protocol definition of ≥ 3 unformed stools per day over 2 consecutive days, a positive C. difficile stool toxin assay, and the requirement of CDI SOC antibiotic therapy, and an adequate clinical response following antibiotic therapy (<3 unformed stools in 24 hours for 2 or more consecutive days).

Cohort 1 Main Exclusion Criteria:

1. Female subjects who are pregnant, breastfeeding, lactating, or planning to become pregnant during the study.
2. Known or suspected toxic megacolon and/or known small bowel ileus.
3. Admitted to or expected to be admitted to an intensive care unit for medical reasons (not just boarding). Note: nursing homes, rehabilitation, assisted living centers and acute care hospitals are acceptable.
4. Absolute neutrophil count of <500 cells/mm^3.
5. Major gastrointestinal surgery (e.g. significant bowel resection or diversion) within 3 months before enrollment (this does not include appendectomy or cholecystectomy), or any history of total colectomy or bariatric surgery (bariatric surgery which does not disrupt the gastrointestinal lumen, i.e., restrictive procedures such as banding, are permitted).
6. History of active inflammatory bowel disease (ulcerative colitis, Crohn's disease, microscopic colitis) with diarrhea believed to be caused by active inflammatory bowel disease in the past 3 months.
7. Concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy (subjects on maintenance chemotherapy may only be enrolled after consultation with the study medical monitor).
8. Any history of fecal microbiota transplantation (FMT) in the past 3 months.

Cohort 2 Main Inclusion Criteria:

1. Subjects 18 years of age or older who had one or more CDI recurrence (as confirmed by a C. difficile stool toxin or PCR test) and have responded to a course of antibiotic treatment.
2. Signed informed consent prior to initiation of any study-specific procedure or treatment. The subject, or their legally authorized representative, must be able to provide written informed consent and understand the potential risks and benefits from study enrollment and treatment.

Cohort 2 Main Exclusion Criteria:

(all Cohort 1 exclusion criteria [#1-8 above] plus the below addition criterion)

9. Previously enrolled in a Seres Therapeutics clinical study. An exception is made for subjects who screened in SERES-012 who did not receive SER-109 and did not previously roll-over to SERES-013.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Wang, MD, Study Director — Seres Therapeutics, Inc.
Locations (97):
- United States (87):
  - (Investigator site), Dothan, Alabama
  - (Investigator site), Sun City West, Arizona
  - (Investigator site), Mather, California
  - (Investigator site), Mountain View, California
  - (Investigator site), Murrieta, California
  - (Investigator site), Northridge, California
  - (Investigator site), Sacramento, California
  - (Investigator site), San Bernardino, California
  - (Investigator site), San Diego, California
  - (Investigator site), San Dimas, California
  - (Investigator site), Simi Valley, California
  - (Investigator site), Thousand Oaks, California
  - (Investigator site), Clearwater, Florida
  - (Investigator site), DeLand, Florida
  - (Investigator site), Hialeah, Florida
  - (Investigator site), Homestead, Florida
  - (Investigator site), Jacksonville, Florida
  - (Investigator site), Miami, Florida
  - (Investigator site), Miami Lakes, Florida
  - (Investigator site), Naples, Florida
  - (Investigator site), Orlando, Florida
  - (Investigator site), Pembroke Pines, Florida
  - (Investigator site), Port Orange, Florida
  - (Investigator site), Athens, Georgia
  - (Investigator site), Atlanta, Georgia
  - (Investigator site), Decatur, Georgia
  - (Investigator site), Marietta, Georgia
  - (Investigator site), Morrow, Georgia
  - (Investigator site), Boise, Idaho
  - (Investigator site), Idaho Falls, Idaho
  - (Investigator site), Chicago, Illinois
  - (Investigator site), Oak Lawn, Illinois
  - (Investigator site), Springfield, Illinois
  - (Investigator site), Evansville, Indiana
  - (Investigator site), Iowa City, Iowa
  - (Investigator site), Kansas City, Kansas
  - (Investigator site), New Orleans, Louisiana
  - (Investigator site), Annapolis, Maryland
  - (Investigator site), Chevy Chase, Maryland
  - (Investigator site), Glen Burnie, Maryland
  - (Investigator site), Boston, Massachusetts
  - (Investigator site), Framingham, Massachusetts
  - (Investigator site), North Dartmouth, Massachusetts
  - (Investigator site), Weymouth, Massachusetts
  - (Investigator site), Worcester, Massachusetts
  - (Investigator site), Chesterfield, Michigan
  - (Investigator site), Detroit, Michigan
  - (Investigator site), Flint, Michigan
  - (Investigator site), Royal Oak, Michigan
  - (Investigator site), Wyoming, Michigan
  - (Investigator site), Rochester, Minnesota
  - (Investigator site), Chesterfield, Missouri
  - (Investigator site), Butte, Montana
  - (Investigator site), Morristown, New Jersey
  - (Investigator site), Neptune City, New Jersey
  - (Investigator site), Buffalo, New York
  - (Investigator site), New York, New York
  - (Investigator site), Charlotte, North Carolina
  - (Investigator site), Greenville, North Carolina
  - (Investigator site), Jacksonville, North Carolina
  - (Investigator site), Kinston, North Carolina
  - (Investigator site), Akron, Ohio
  - (Investigator site), Centerville, Ohio
  - (Investigator site), Cincinnati, Ohio
  - (Investigator site), Cleveland, Ohio
  - (Investigator site), Mentor, Ohio
  - (Investigator site), Toledo, Ohio
  - (Investigator site), Camp Hill, Pennsylvania
  - (Investigator site), Harrisburg, Pennsylvania
  - (Investigator site), Pittsburgh, Pennsylvania
  - (Investigator site), Sayre, Pennsylvania
  - (Investigator site), Providence, Rhode Island
  - (Investigator site), Union City, Tennessee
  - (Investigator site), Cypress, Texas
  - (Investigator site), Garland, Texas
  - (Investigator site), Houston, Texas
  - (Investigator site), McKinney, Texas
  - (Investigator site), Pasadena, Texas
  - (Investigator site), San Antonio, Texas
  - (Investigator site), Southlake, Texas
  - (Investigator site), Spring, Texas
  - (Investigator site), Ogden, Utah
  - (Investigator site), Riverton, Utah
  - (Investigator site), Salt Lake City, Utah
  - (Investigator site), Spokane, Washington
  - (Investigator site), Tacoma, Washington
  - (Investigator site), Milwaukee, Wisconsin
- Canada (10):
  - (Investigator site), Calgary, Alberta
  - (Investigator site), Vancouver, British Columbia
  - (Investigator site), Victoria, British Columbia
  - (Investigator site), St. John's, Newfoundland and Labrador
  - (Investigator site), London, Ontario
  - (Investigator site), North Bay, Ontario
  - (Investigator site), Scarborough Village, Ontario
  - (Investigator site), Chicoutimi, Quebec
  - (Investigator site), Québec, Quebec
  - (Investigator site), Sainte-Foy, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kraft CS, Sims M, Silverman M, Louie TJ, Feuerstadt P, Huang ES, Khanna S, Berenson CS, Wang EEL, Cohen SH, Korman L, Lee C, Kelly CR, Odio A, Cook PP, Lashner B, Ramesh M, Kumar P, De A, Memisoglu A, Lombardi DA, Hasson BR, McGovern BH, von Moltke L, Pardi DS; ECOSPOR III and ECOSPOR IV investigators. Integrated Safety and Efficacy Analyses of Phase 3 Trials of a Microbiome Therapeutic for Recurrent CDI. Infect Dis Ther. 2024 Oct;13(10):2105-2121. doi: 10.1007/s40121-024-01007-z. Epub 2024 Jun 28. PMID 38941068
- [Derived] Sims MD, Khanna S, Feuerstadt P, Louie TJ, Kelly CR, Huang ES, Hohmann EL, Wang EEL, Oneto C, Cohen SH, Berenson CS, Korman L, Lee C, Lashner B, Kraft CS, Ramesh M, Silverman M, Pardi DS, De A, Memisoglu A, Lombardi DA, Hasson BR, McGovern BH, von Moltke L; ECOSPOR IV Investigators. Safety and Tolerability of SER-109 as an Investigational Microbiome Therapeutic in Adults With Recurrent Clostridioides difficile Infection: A Phase 3, Open-Label, Single-Arm Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2255758. doi: 10.1001/jamanetworkopen.2022.55758. PMID 36780159

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Overall, there were 64 sites in the United States and 8 sites in Canada that enrolled participants between 2017 to 2021.
Groups:
- Cohort 1: Rollover participants from study SERES-012, who received oral dose of SER-109 in 4 capsules once daily for 3 consecutive days in SERES-013 study.
- Cohort 2: Newly enrolled participants who received oral dose of SER-109 in 4 capsules once daily for 3 consecutive days.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 29 | 234
Completed 8-week Follow-up | 29 | 228
Completed (Completed 24-week Follow-up) | 27 | 222
Not Completed | 2 | 12
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Death | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 29 | 234 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.7 (12.46) | 63.1 (15.79) | 64.0 (15.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 162 | 180
  Male | 11 | 72 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 29 | 214 | 243
  Black or African American | 0 | 14 | 14
  Asian | 0 | 5 | 5
  American Indian or Alaska Native | 0 | 1 | 1
  Not Hispanic or Latino | 29 | 214 | 243
  Hispanic or Latino | 0 | 20 | 20
Antibiotic regimen for qualifying episode [Count of Participants; unit: Participants]
  Vancomycin | 22 | 169 | 191
  Fidaxomicin | 7 | 65 | 72

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Recurrence of CDI and Sustained Clinical Response
Description: Cohort 1: Recurrence of CDI up to 8 Weeks after treatment. Recurrence was determined by stool Clostridioides difficile toxin assay. Sustained clinical response was the absence of CDI recurrence up to 8 Weeks after treatment.
Time Frame: Up to Week 8
Population: The analysis population consisted of all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 29
Participants
  Number of participants with CDI recurrence | 4
  Number of participants with sustained response | 25

2. Primary Outcome: Cohort 2: Recurrence of CDI and Sustained Clinical Response
Description: Cohort 2: Recurrence of CDI up to 8 and 12 Weeks after treatment. Recurrence was determined by stool Clostridioides difficile toxin assay. Sustained clinical response was the absence of CDI recurrence up to 8 and 12 Weeks after treatment.
Time Frame: Up to Weeks 8 and 12
Population: The analysis population consisted of all enrolled participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 2
Number analyzed (Participants) | 234
Participants
  Week 8: Number of participants with CDI recurrence | 19
  Week 8: Number of participants with sustained clinical response | 215
  Week 12: Number of participants with CDI recurrence | 23
  Week 12: Number of participants with sustained clinical response | 211

ADVERSE EVENTS:
Time Frame: 24 weeks follow-up starting Day 1 post-dosing with SER-109
Description: All adverse events were collected from Day 1 post-dosing to Week 8. From Week 8 onwards to the end of study (Week 24), only serious adverse events and adverse events of special interest (e.g., invasive infections) were collected.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/29 | 8/234
Serious Adverse Events (participants affected / at risk) | 1/29 | 32/234
Other Adverse Events (participants affected / at risk) | 14/29 | 68/234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=29) | Cohort 2 (N=234)
Cellulitis (Infections and infestations) | 0 | 4
Urinary tract infection (Infections and infestations) | 0 | 3
Clostridium difficile colitis (Gastrointestinal disorders) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 4
Corona virus infection (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Cytomegalovirus viremia (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 0 | 1
Escherichia bacteremia (Infections and infestations) | 0 | 1
Necrotizing fasciitis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2
Ascites (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric volvulus (Gastrointestinal disorders) | 0 | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Facial paralysis (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2
End stage renal disease (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Amylase increased (Investigations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Chest wall hematoma (Musculoskeletal and connective tissue disorders) | 0 | 1
Chronic recurrent multifocal osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Death due to natural causes (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Device occlusion (Product Issues) | 0 | 1
Vasculitic ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=29) | Cohort 2 (N=234)
Diarrhea (Gastrointestinal disorders) | 10 | 48
Flatulence (Gastrointestinal disorders) | 4 | 16
Nausea (Gastrointestinal disorders) | 3 | 17
Abdominal pain (Gastrointestinal disorders) | 3 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT03183141/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT03183141/SAP_001.pdf